CLINICAL TRIAL: NCT05236985
Title: Randomized Double-Blinded Clinical Trial of Oxytocin Bolus Versus Infusion in Elective Cesarean Section
Brief Title: Oxytocin Bolus Versus Infusion in Elective Cesarean Section"
Acronym: INBOX
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Stony Brook University (Other)
Responsible Party: Principal Investigator, Tiffany E. Angelo, D.O., Assistant Professor Division Chief: Women's Anesthesiology, Stony Brook University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Other
Other Study IDs: IRB 2021-00558
Record Dates: First submitted 2021-12-23; First posted 2022-02-11 (Actual); Last update posted 2024-03-15 (Actual); Status verified 2024-03

CONDITIONS: Elective Cesarean Section
Keywords: Oxytocin, bolus, infusion

STUDY DESIGN:
Intervention Model Description: Randomized, double-blinded, 2-arm, parallel study.
Who Masked: Participant, Care Provider, Investigator
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Bolus arm (Active Comparator): Patients will receive 3 IU oxytocin IV bolus over 15 seconds after delivery of the baby/uterine cord clamping and a maintenance infusion of 0.9% Saline will be started at 225ml/hr. If uterine tone is inadequate after 3 minutes, a second bolus of 3 IU oxytocin will be given. If uterine tone is inadequate after an additional 3 minutes, a third bolus of 3 IU Oxytocin IV is given over 15 seconds. If after an additional 3 mins uterine tone is still inadequate, a second infusion consisting of oxytocin 3 IU/hr is started at 100ml/hrs and continued for a total of 4 hours, second line uterotonic agents (Methergine, Hemabate and/ or Cytotec) will be given, and the maintenance 0.9% Saline infusion will be changed to 450 ml/hr for a total of 1 hour, then changed to 38 ml/ hour for the following 3 hours. If uterine tone is considered adequate at 3, 6 or 9 minutes, a second infusion of oxytocin 3 IU/hr (100ml/hr) is started and maintained for 4 hours.
  Interventions: Drug: Oxytocin bolus or oxytocin infusion
- Infusion arm (Active Comparator): Patients will receive a bolus of IV 0.9% Saline over 15 seconds after delivery of the baby/uterine cord clamping and a maintenance infusion of 18 IU/hr Oxytocin IV (225ml/hr). If uterine tone is inadequate after 3 minutes, a second bolus of 0.9% Saline will be given. If uterine tone is inadequate after another 3 minutes, a third bolus of 0.9% Saline will be given. If after another 3 mins uterine tone is inadequate, a second infusion of 0.9% Saline will be started for 4 hours, second line uterotonic agents (Methergine, Hemabate and/or Cytotec) will be given, and the Oxytocin infusion will be changed to 36 IU/hour (450 ml/hr) for a total of 1 hour, and then changed to 38 ml/hr for the following 3 hours. If uterine tone is considered adequate at 3, 6 or 9 minutes, a second infusion of 0.9% Saline at 100 ml/hr will be started and maintained for 4 hours, along with the maintenance infusion of 18 IU/hr (225 ml/ hr) for a total of 1 hour, then changed to 38 ml/hr for an additional 3 hours.
  Interventions: Drug: Oxytocin bolus or oxytocin infusion

INTERVENTIONS:
Drug: Oxytocin bolus or oxytocin infusion — On the day of surgery, the patients will be randomized to either bolus or infusion administration of oxytocin.
  On the day of the procedure, periprocedural data and patient satisfaction (single question) will be recorded.

SUMMARY:
Bolus administration of oxytocin is superior to infusion in time to achieving adequate uterine tone.

DETAILED DESCRIPTION:
Oxytocin is the most commonly used uterotonic agent worldwide to achieve adequate uterine tone and prevent postpartum hemorrhage. Over the past decade, the trend has been towards lowering the dose to reduce oxytocin-related adverse effects including nausea, hypotension, chest pain, EKG changes, and maternal death. However, the optimal strategy for oxytocin administration remains controversial. Prior literature found bolus doses less than 5 IU to be effective in achieving adequate uterine tone with a significant reduction in adverse side effects. There is limited high quality data comparing bolus versus infusion administration of oxytocin. The current standard of care at the institution is an infusion of oxytocin 18 IU/hour (0.3 IU/min) and has been proven to be effective in achieving adequate uterine tone. However, the time to uterine tone appears to be slightly longer (3-4 mins) with the infusion method. Given that the estimated uterine blood flow is between 500-700 mls/min, the uterus can lose a significant amount of blood per second if uterine tone is not achieved quickly. Thus, the purpose of this research study is to compare bolus and infusion administration of oxytocin on parturients undergoing elective cesarean section. The primary objective of this study is to test the hypothesis that administration by bolus (vs. standard of care infusion) results in more rapid achievement of adequate uterine tone. Secondary objectives include determining estimated blood loss, prevalence of hypotension, nausea, vomiting, and patient satisfaction.

ELIGIBILITY:
Inclusion Criteria:

* Parturients between the ages of 18 to 45 with singleton pregnancies
* Undergoing elective cesarean section under spinal anesthesia
* American Society of Anesthesia (ASA) physical status class I or II
* Patients must be able to provide written informed consent

Exclusion Criteria:

* Parturients in labor or ruptured membranes
* Multiple gestation
* Risk factors predisposing to uterine atony (history of placenta previa, preeclampsia, diabetes mellitus macrosomia, hydramnios, bleeding diathesis, uterine fibroids)
* History of uterine atony or postpartum hemorrhage
* History of inherited or acquired coagulation disorders, thrombocytopenia (platelet count <100), or anemia (hemoglobin < 8)
* History of allergy to oxytocin
* Patients not alert and orientated to person, place, and date. Patient must have, in the investigator's opinion, the physical and mental capacity to answer survey questions

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — Pregnant women
Enrollment: 120 (Estimated)
Dates: Start 2022-03-15 (Actual); Primary Completion 2024-12-15 (Estimated); Study Completion 2024-12-15 (Estimated)

PRIMARY OUTCOMES:
Number/Proportion of Participants with Adequate Uterine tone | 2 minutes
  Adequacy of uterine tone (yes/no) at 2 minutes after the baby is born/umbilical cord clamped.

SECONDARY OUTCOMES:
Patient satisfaction questionnaire (Scale 0 to 10, 0 being complete dissatisfaction and 10 being highly satisfied | 2± 1 hours after surgery
  Patients will complete a questionnaire 2± 1 hours after surgery

CONTACTS AND LOCATIONS:
Overall Officials: Tiffany E Angelo, DO, Principal Investigator — Stony Brook University
Locations (1):
- Stony Brook University, Stony Brook, New York, United States

IPD SHARING:
Plan to Share IPD: No
Data will not be shared

REFERENCES:
- [Background] Say L, Chou D, Gemmill A, Tuncalp O, Moller AB, Daniels J, Gulmezoglu AM, Temmerman M, Alkema L. Global causes of maternal death: a WHO systematic analysis. Lancet Glob Health. 2014 Jun;2(6):e323-33. doi: 10.1016/S2214-109X(14)70227-X. Epub 2014 May 5. PMID 25103301
- [Background] Balki M, Tsen L. Oxytocin protocols for cesarean delivery. Int Anesthesiol Clin. 2014 Spring;52(2):48-66. doi: 10.1097/AIA.0000000000000016. No abstract available. PMID 24667448
- [Background] Terblanche N, Otahal P, Messmer A, Wright P, Patel S, Nathan K, Sharman JE. An observational cohort study of 3 units versus 5 units slow intravenous bolus oxytocin in women undergoing elective caesarean delivery. J Physiol Pharmacol. 2017 Aug;68(4):547-553. PMID 29151071
- [Background] Fuchs AR, Fuchs F, Husslein P, Soloff MS. Oxytocin receptors in the human uterus during pregnancy and parturition. Am J Obstet Gynecol. 1984 Nov 15;150(6):734-41. doi: 10.1016/0002-9378(84)90677-x. PMID 6093538
- [Background] Joseph J, George SK, Daniel M, Ranjan RV. A randomised double-blind trial of minimal bolus doses of oxytocin for elective caesarean section under spinal anaesthesia: Optimal or not? Indian J Anaesth. 2020 Nov;64(11):960-964. doi: 10.4103/ija.IJA_377_20. Epub 2020 Nov 1. PMID 33487681